CLINICAL TRIAL: NCT06945146
Title: The Comprehensive Assessment of BCR-ABL1 Gene Expression and Genetic Variations by qRT-PCR and NGS Assays in Chronic Myeloid Leukemia Patients Who Are Treated With Ponatinib (CAP Study)
Brief Title: Genomics Study in CML Patients With Ponatinib Treatment
Acronym: CAP
Status: Completed | Type: Observational
Sponsor: Dong-Wook Kim (Other)
Collaborators: Ulsan National Institute of Science and Technology (Unknown); Takeda (Industry)
Responsible Party: Sponsor-Investigator, Dong-Wook Kim, professor, Eulji University Hospital
Organization: Eulji University Hospital (Other)
Other Study IDs: KC20MISI0507
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-12

CONDITIONS: Chronic Myelogenous Leukemia, BCR-ABL1 Positive
Keywords: ponatinib; tyrosine kinase inhibitor; resistance; intolerance; genetic variation; next generation sequencing
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- CML patients failed to TKIs except Ponatinib: The study will involve 100 patients with BCR-ABL1-positive CML who failed to prior targeted therapy other than ponatinib. Patients receiving ponatinib 45 mg once daily as a second-line or later therapy will be enrolled.
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Ponatinib treatment will be initiated per usual treatment procedure at 45 mg once daily p.o., which will be gradually decreased to 30 mg and 15 mg according to the predefined criteria based on responsiveness to treatment and AEs in the course of the treatment.
  Other Names: Iclusig

SUMMARY:
This study will evaluate whether responsiveness and adverse events (AEs) to second-line or later ponatinib treatment are associated with genetic variations as measured by real-time quantitative polymerase chain reaction (qRT-PCR) and next-generation sequencing (NGS) in patients with CML of any stage who failed prior multiple targeted therapies except ponatinib.

DETAILED DESCRIPTION:
Ponatinib treatment will be initiated per usual treatment procedure at 45 mg once daily p.o., which will be gradually decreased to 30 mg and 15 mg according to the predefined criteria based on responsiveness to treatment and AEs in the course of the treatment. A total of 100 subjects will be enrolled within 24 months after the first subject enrollment, and ponatinib treatment will continue for 24 months after the initial dosing of ponatinib in each enrolled subject. Routine ponatinib treatment will continue at the investigator's discretion until disease progression, the occurrence of unacceptable toxicity, subject's withdrawal of consent, or occurrence of any reason for discontinuation specified in the protocol.

All molecular analysis samples will be collected, transferred, and managed by the Catholic Leukemia Research Institute, and NGS will be performed.

<Eligibility>

1. Adults with BCR-ABL1-positive CML
2. Subjects who were resistant or intolerant to prior targeted therapy other than ponatinib and with an indication for ponatinib treatment according to the acceptance criteria by the Ministry of Food and Drug Safety (MFDS)
3. Women of childbearing potential (WOCBP) should have a negative serum or urine pregnancy test (with a sensitivity of at least 25 IU/L or equivalent to HCG) within 24 hours before initiating ponatinib treatment
4. Written informed consent to ponatinib treatment

<Outcome Measures>

1. Primary endpoint

   - 24 months dynamics of BCR-ABL1 gene expression by qRT-PCR
2. Secondary endpoints

   * Type and frequency of novel genetic variations (mutations, gene expressions, CNV, INDEL, etc.)
   * Cobll1/GCA/novel gene network identification: functional tests using Western blot/Knock-down assay
3. Safety endpoints : To explore the dynamics of adverse events according to dose changes up to 24 months

   * Frequency and severity of skin rash, fever, hypertension, pancreatitis and vascular events as common adverse events
   * Frequency and severity of rare adverse events
   * Treatment intolerance is defined as recurrence of a Grade ≥3 hematologic AE, or a Grade ≥2 non-hematologic AE requiring permanent discontinuation of ponatinib per protocol despite dose reduction

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to and capable of providing informed consent
* Adults with BCR-ABL1-positive CML

  1. Males and females aged 18 years and above
  2. Adequate organ function
* Subjects who were resistant or intolerant to prior targeted therapy other than ponatinib and with an indication for ponatinib treatment according to the acceptance criteria by the Ministry of Food and Drug Safety (MFDS)
* Women of childbearing potential (WOCBP) should have a negative serum or urine pregnancy test (with a sensitivity of at least 25 IU/L or equivalent to HCG) within 24 hours before initiating ponatinib treatment
* Female subjects who are not breastfeeding

Exclusion Criteria:

* Patients who were previously treated with ponatinib
* Patients aged below 18 years of age
* Diagnosis of severe comorbidity at baseline
* Any other cancers within 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve 100 patients with BCR-ABL1-positive CML who failed to prior targeted therapy other than ponatinib. Patients receiving ponatinib 45 mg once daily as a second-line or later therapy will be enrolled.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Dynamics of BCR-ABL1 gene expression by qRT-PCR | 24 months
  To explore the dynamics of BCR-ABL1 kinetics by Ponatinib

SECONDARY OUTCOMES:
Type and frequency of novel genetic variations (mutations, gene expressions, CNV, INDEL, etc.) | 24 months
  To explore the dynamics of various genetic variations in Ponatinib failed patients
Cobll1/GCA/novel gene network identification: functional tests using Western blot/Knock-down assay | 24 months
  To identify novel genetic networks in Ponatinib failed patients

OTHER OUTCOMES:
Frequency and severity of skin rash, fever, hypertension, pancreatitis and vascular events as common adverse events and Frequency and severity of rare adverse events | 24 months
  To explore the dynamics of adverse events according to dose changes up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wook Kim, MD, PhD, Principal Investigator — Eulji University
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided